CLINICAL TRIAL: NCT04535830
Title: The Effectiveness of Flash Glucose Monitoring System on Glycemic Control in Patients With New-onset Type 2 Diabetes#A Randomized Controlled Trial
Brief Title: The Effectiveness of Flash Glucose Monitoring System on Glycemic Control in Patients With New-onset Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yufan Wang, Director of endocrinology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0304N18020
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2; Flash Glucose Monitoring
Keywords: type 2 diabetes; Glucose management; Flash glucose monitoring system
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized controlled trial. The investigators plan to recruit 200 persons with type 2 diabetes diagnosed within six months. Participants will be randomly assigned (1:1) to either use of a flash glucose monitoring system(FSL) or self-monitoring blood glucose(SMBG) . All participants need to wear the flash glucose monitoring sensor at baseline and at the end of the experiment for data analysis.During the three months of experiment,participants at the FSL group will wear a flash glucose monitoring sensor for 14 days and have a care visit every month,while people at SMBG group will monitor their glucose by pricking a finger at home and receive a care visit every month as well.
  The primary outcome is the between-group difference in mean HbA1c at 3 months. Meanwhile,researchers want to know whether differences in glucose variability and diabetes-specific distress between two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flash glucose monitor system(FSL) (Experimental): Except at baseline and at the end of the experiment,participants at the FSL group will be asked to wear a flash glucose monitoring sensor for a period of 2 weeks and have a care visit every month.
  Interventions: Device: Flash Glucose Monitoring System
- Self-monitoring blood glucose(SMBG) (No Intervention): People at SMBG group will wear the sensor at baseline and at the end of the experiment for data analysis only,and will have a care visit every month.

INTERVENTIONS:
Device: Flash Glucose Monitoring System — During the three months experimental period,participants at the FSL group will be asked to wear a flash glucose monitoring sensor for a period of 2 weeks and have a care visit every month while people at SMBG group will receive a care visit every month.
  Other Names: Freestyle Libre
  Arms: Flash glucose monitor system(FSL)

SUMMARY:
The purpose of this study is to determine if Flash glucose monitoring system improves glycemic control in adults with new-onset type 2 diabetes

DETAILED DESCRIPTION:
People with new-onset type 2 diabetes who achieve and sustain glycemic targets is important for reducing the risk of complications and all-cause mortality.Glucose monitoring is the key point of diabetes management.Continuous glucose monitoring(CGM)can identify day-to-day glucose profiles to guide management decisions.Flash glucose monitoring is a variant of CGM and is factory calibrated,requiring no finger pricks.The purpose of this study is to determine if Flash glucose monitoring improves glycemic control in adults with new-onset type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* peolpe with type 2 diabetes in accordance with the dignosed criteria of CDS2017
* type 2 diabetes duration of <6months
* with certain read-write ability
* willing to use FSL or follow study protocol

Exclusion Criteria:

* acute complication of diabetes condition(DKA,HHH)
* pregnancy,lactating or planning pregnancy
* allergy to adhesive tape
* skin with large area of rubefaction and wounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
the between-group difference in mean HbA1c | 3months
  difference in mean HbA1c between FSL group and SMBG group

SECONDARY OUTCOMES:
the between-group difference in mean time in target glucose range | 3months
  difference in mean time in target glucose range between FSL group and SMBG group
the between-group difference in mean time in hypoglycemia | 3months
  difference in mean time in hypoglycemia between FSL group and SMBG group
the between-group difference in mean time in other biochemical indexes,such as LDL-C,TC,TG and so on | 3months
  difference in some biochemical indexes between FSL group and SMBG group

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China